CLINICAL TRIAL: NCT00708812
Title: Paclitaxel Plus Carboplatin (TC) Versus TC Plus Endostar in Patients With Advanced Non-small Cell Lung Cancer(NSCLC): a Randomized, Double-blind, Placebo-controlled, Multicentre Study
Brief Title: Paclitaxel Plus Carboplatin With or Without Endostar in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Simcere-Medgenn Bio-pharmaceutical Co., Ltd (Industry)
Responsible Party: Jinsheng Ren, Shandong Simcere-Medgenn Bio-pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XYL014
Record Dates: First submitted 2008-06-21; First posted 2008-07-02 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Endostar; Paclitaxel; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — CP protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The control group (Active Comparator): paclitaxel-carboplatin
  Interventions: Drug: paclitaxel-carboplatin
- The treatment group (Experimental): paclitaxel-carboplatin plus Endostar
  Interventions: Drug: Endostar(Recombinant Human Endostatin Injection); Drug: paclitaxel-carboplatin

INTERVENTIONS:
Drug: Endostar(Recombinant Human Endostatin Injection) — Endostar 7.5mg/m2 on d8-d21 in each 21-day cycle
  Arms: The treatment group
Drug: paclitaxel-carboplatin — paclitaxel, 175mg/m2, iv, d1, q3w; carboplatin, AUC 5, iv, d1, q3w

SUMMARY:
In this randomized, double-blind, placebo-controlled, multicentre trial, 126 patients between July 5, 2007 and July 30, 2008 were enrolled from 10 centers. The leader units are Shanghai Chest Hospital Affiliated to Shanghai Jiao-Tong University and Shanghai Changzheng Hospital. All eligible patients received 1 cycle (21 days) of TC chemotherapy. After chemotherapy, patients evaluated as SD (Stable Disease) or above were randomized to receive endostar plus TC or TC alone for 3 cycles, 21 days as one cycle.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed, previously untreated stage IIIB or IV NSCLC
* age of 18-75 years
* at least one measurable lesion (RECIST)
* patients evaluated as SD or above after 1 cycle (21 days) of TC chemotherapy .
* adequate hematologic, cardiac, renal, and hepatic function
* ECOG PS 0-2

Exclusion Criteria:

* symptomatic brain metastases
* bone metastases with complications
* major organ dysfunction
* bleeding diathesis or coagulopathy
* pregnant or lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | every 2 months until disease progression

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | the end of each cycle
Overall Survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China